CLINICAL TRIAL: NCT04725448
Title: A Single-arm Exploratory Clinical Study on the Efficacy and Safety of Toripalimab Combined With Bevacizumab, Nab-paclitaxel and Carboplatin for Untreated Metastatic Pulmonary Sarcomatoid Carcinoma
Brief Title: Toripalimab Combined With Bevacizumab, Nab-paclitaxel and Carboplatin for Untreated Metastatic Pulmonary Sarcomatoid Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sichuan Cancer Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Juan LI, MD, MD, Sichuan Cancer Hospital and Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS001-ISS-CO200
Record Dates: First submitted 2021-01-06; First posted 2021-01-26 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Pulmonary Sarcomatoid Carcinoma; Non-small Cell Lung Cancer; Lung Diseases; Thoracic Neoplasms
Keywords: PSC; NSCLC; Toripalimab; immunity therapy; Anti-angiogenesis; Platinum-containing dual-agent chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Diseases; Thoracic Neoplasms | interventions — toripalimab; Bevacizumab; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Toripalimab Combined With Bevacizumab, Nab-paclitaxel and Carboplatin (Experimental): Drugs: Toripalimab, 240mg (6ml)/bottle, ivgtt, d1, q3w, administration until PD or death, the longest use time is two years.
  Drugs: Bevacizumab, 7.5mg/kg, ivgtt, d1, q3w,the longest use time is two years.
  Drugs: Nab-paclitaxel, 260mg/m2,ivgtt,d1 or 130mg/m2,ivgtt,d1,8, q3w, up to six cycles.
  Drugs: Carboplatin, AUC=4～5, ivgtt, d1, q3w, up to six cycles.
  Interventions: Drug: Toripalimab; Drug: Bevacizumab; Drug: Nab-paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Toripalimab — 240mg, ivgtt, d1, every 3 weeks until disease progress or intolerable toxicity, up to 2 years of administration
  Other Names: JS001; Toripalimab Injection; TuoYI; Teruipuli Dankang
Drug: Bevacizumab — 7.5mg/kg, ivgtt, d1, every 3 weeks, up to 2 years of administration
  Other Names: Bevacizumab Injection; Avastin; Bei Fa Zhu Dankang Zhusheye
Drug: Nab-paclitaxel — 260mg/m2,d1 or 130mg/m2,d1,8, ivgtt, every 3 weeks, up to 6 cycles
  Other Names: ABRAXANE; paclitaxel protein-bound particles for injectable suspension
Drug: Carboplatin — AUC=4～5, d1, ivgtt, every 3 weeks, up to 6 cycles
  Other Names: Carboplatin injection

SUMMARY:
This study aimed to evaluate the efficacy and safety of first-line Toripalimab combined with bevacizumab, nab-paclitaxel and carboplatin in the treatment of patients with advanced pulmonary sarcomatoid carcinoma.

DETAILED DESCRIPTION:
Pulmonary sarcomatoid carcinoma(PSC) is a rare primary lung cancer, which belongs to the category of non-small cell lung cancer(NSCLC), accounting for about 0.3%-1.3% of lung cancers .Platinum-based combination chemotherapy is the standard adjuvant chemotherapy and palliative chemotherapy for NSCLC, and it is also commonly used for PSC. Advanced PSC has a low response rate to systemic chemotherapy and a short duration of curative effect. The primary progression rate of aggressive platinum-based chemotherapy is 60%-70%, showing that PSC is highly resistant to multiple chemotherapeutics. In recent years, the progress of targeting MET tyrosine kinase mutations has been relatively rapid, but most of the mutant PSCs targeting EGFR, KRAS, ALK, and BRAF V600E are case reports and there is no effective treatments. Immunotherapy has rewritten the treatment pattern of NSCLC. However, the current application of immunotherapy in PSC are mostly case reports. In immunotherapy, IMpower150 research data suggests that the combination of immunity and anti-angiogenesis + platinum-containing dual-agent chemotherapy can bring sustained OS benefits in NSCLC patients , and safety tolerated. However, PSC has moderate to high tumor mutation burden (TMB >10 mutations/Mb). This high mutation rate may increase tumor immunogenicity, making immunotherapy a better treatment option. At the same time, VEGF, as a cytokine that promotes the growth and differentiation of vascular endothelial cells, plays a decisive role in promoting tumor neovascularization. In this regard, immunotherapy combined with anti-angiogenesis and chemotherapy is worth exploring in the treatment of PSC.

ELIGIBILITY:
Inclusion Criteria:

* 1.18 to 75 years old, no gender limit;
* 2.ECOG PS: 0～2 points;
* 3.Untreated patients with stage IV pulmonary sarcomatoid carcinoma are staged according to the AJCC eighth edition non-small cell lung cancer staging standard;
* 4.Pulmonary sarcomatoid carcinoma confirmed by histopathology has at least one measurable lesion according to RECIST standard 1.1, and the lesion has not received radiotherapy;
* 5.The functions of important organs meet the following requirements (no blood components and cell growth factors are allowed to be used 2 weeks before the start of the research treatment) : Absolute Neutrophil Count (ANC) ≥1.5×10 E+9/L, Hemoglobin (HB) ≥9g/dL, Platelets (PLT)≥90×10 E+9/L, Serum Albumin (ALB)≥2.8g/dL, Total Bilirubin (TBIL) ≤1.5 ULN, ALT、AST≤2.5 UILN(If abnormal liver function is caused by liver metastasis, ≤5 ULN), Serum creatinine sCr≤1.5 ULN, endogenous creatinine clearance ≥50ml/min (Cockcroft-Gault formula) ,Normal thyroid function;
* 6.Expected survival time ≥ 3 months;
* 7.Female subjects with fertility should undergo a urine or serum pregnancy test within 72 hours before receiving the first study drug administration, and prove to be negative, and are willing to use effective during the test period to 3 months after the last administration Methods of contraception. For male subjects whose partners are women of childbearing age, effective methods of contraception should be used during the trial and within 3 months after the last administration;
* 8.The patients joined the study voluntarily and signed an informed consent form (ICF). They had good compliance and cooperated with follow-up.

Exclusion Criteria:

* 1.Patients with pathological types and primary lesions that do not meet the inclusion criteria;
* 2.There is known evidence that patients have mutations in any of the genes above EGFR, ROS-1, ALK, and c-MET;
* 3.Suffer from any active autoimmune diseases, such as interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism (can be included after hormone replacement therapy is normal);
* 4.Known to be allergic to other monoclonal macromolecular protein preparations, or to any of the components of Toripalimab;
* 5.Have received other PD-1 monoclonal antibody therapy or other immunotherapy against PD-1/PD-L1;
* 6.Active infection or fever of unknown origin occurred during the screening period and before the first administration>38.5℃ (according to the judgment of the investigator, the subject can be included in the group for fever caused by the tumor);
* 7.Suffering from uncontrolled clinical symptoms or diseases of the heart, such as: (1) Heart failure above NYHA II; (2) Unstable angina pectoris; (3) Myocardial infarction occurred within 1 year; (4) Patients with clinically significant supraventricular or ventricular arrhythmia requiring clinical intervention.
* 8.Suffering from high blood pressure and cannot be well controlled by antihypertensive drugs (systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 100 mmHg);
* 9.Abnormal coagulation function (INR>2.0, PT>16s), have bleeding tendency or are receiving thrombolytic therapy, and allow preventive use of low-dose aspirin and low-molecular-weight heparin;
* 10.Obvious coughing up blood or hemoptysis of 10ml or more per day in the 2 months before enrollment;
* 11.Have significant clinically significant bleeding symptoms or have a clear bleeding tendency within 3 months before enrollment;
* 12.Suffer from congenital or acquired immune function defects (such as HIV infection);
* 13.Received anti-tumor monoclonal antibody (mAb) within 4 weeks before the first use of the study drug, or the adverse event caused by the previously received drug has not recovered (ie ≤ grade 1 or reached the baseline level). Note: Except for subjects with ≤ Grade 2 neuropathy or ≤ Grade 2 hair loss, if the subject has undergone major surgery, the toxic reaction and/or complications caused by the surgical intervention must be fully recovered before starting treatment;
* 14.Live vaccines have been vaccinated within 4 weeks before the first use of the study drug. Inactivated virus vaccines for seasonal influenza and injection are allowed, but live attenuated influenza vaccines for nasal use are not allowed;
* 15.According to the judgment of the investigator, the subject has other factors that may cause him to be forced to terminate the study halfway, such as suffering from other serious diseases (including mental illness) requiring combined treatment, severely abnormal laboratory test values, family or social factors, It may affect the safety of subjects or the collection of experimental data;
* 16.The investigator judged other situations not suitable for inclusion in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2021-04-06 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Progress Free Survival(PFS) | up to 2 years
  It is defined as the time interval from randomization of patients to disease progression or death, whichever comes first. There was no progress or the time of disease progression was not recorded when the trial was withdrawn, and the date of the last examination was used as the end date.

SECONDARY OUTCOMES:
Overall response rate(ORR) | up to 2 years
  The proportion of patients with a best overall confirmed response of CR or PR in the whole body as assessed per RECIST 1.1 by the investigator.
Disease Control Rate(DCR) | up to 2 years
  The proportion of patients with a best overall response of CR, PR or SD in the whole body, as assessed per RECIST 1.1 by the investigator.
Overall Survival(OS) | up to 2 years
  Defined as the time interval from randomization to death. If the patient continues to survive or his life or death is unknown, the date of death will be reviewed using the latest point in time when the patient is still alive.
Incidence of AEs | up to 2 years
  AEs per Common Terminology Criteria for Adverse Events (CTCAE V5.0)
the quality of life (QoL) | up to 2 years
  Analysis of changes from baseline using the quality of life (QoL) instrument

CONTACTS AND LOCATIONS:
Overall Officials: Juan Li, MD, Principal Investigator — Sichuan Cancer Hospital and Research Institute
Locations (1):
- Sichuan Cancer Hospital, Chengdu, Sichuan/China, China

IPD SHARING:
Plan to Share IPD: No